CLINICAL TRIAL: NCT05074043
Title: COVID-19 Associated Mucormycosis: A Multidisciplinary Dilemma in Assiut University Hospital
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa mahmoud Abd El Rady, lecturer, Assiut University
Other Study IDs: COVID-19 with mucormycosis
Record Dates: First submitted 2021-10-05; First posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Mucormycosis
MeSH Terms: conditions — Mucormycosis | interventions — Antiviral Agents; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- covid19: covid 19 proven by clinical, PCR. not associated with mucor
- covid19 associated with mucor: covid19 associated with mucor proven by clinical, histopathological
  Interventions: Combination Product: antiviral, surgical

INTERVENTIONS:
Combination Product: antiviral, surgical — surgical debridment
  Groups: covid19 associated with mucor

SUMMARY:
We aimed to describe the frequency; presentations, predictors, in-hospital outcome of mucormycosis patients in the scope of COVID-19.

All patients with COVID-19 associated Mucormycosis (CAM) admitted to Assuit University Hospital between March 1, 2021, and July 30, 2021, were included in this study. The patient characteristics, the site of mucormycosis, the comorbidities, the steroids usage, and the outcome were analyzed in people with COVID-19.

ELIGIBILITY:
Inclusion Criteria:We recruited all cases admitted to Assuit University Hospital for the management of COVID-19 and/or associated complications between March 1, 2021, and July 30, 2021, specifically those with probable mucormycosis based on clinical condition. At various times, internists, intensivists, neurologists, and otolaryngologists were among the specialists who assessed and treated them. Clinical; radiological and histopathological confirmed cases of mucormycosis with coexisting or previous history of COVID-19 were included in this study.

-

Exclusion Criteria:Participants with fungal infections other than mucormycosis or without a confirmed diagnosis of COVID-19 (or serological evidence of preceding COVID-19) were excluded.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with mucormycosis in a confirmed diagnosis of COVID-19
Sampling Method: Probability Sample
Enrollment: 433 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
incidence of covid19 associated mucor | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Marwa Abdelrady, Asyut, Egypt